CLINICAL TRIAL: NCT01241656
Title: Acceleration Adoption of Comparative Effectiveness Research Results With Patient Decision Support Intervention and Treatment (DESI)- Study 1
Brief Title: Decision Support Interventions (DESI) for Prostate Cancer Screening - Study 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Palo Alto Medical Foundation (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Carmen Lewis, MD, MPH, Associate Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 10-1317; 1R18AE000023-01 (NIH)
Record Dates: First submitted 2010-11-15; First posted 2010-11-16 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Healthy Men Age 50 Who Are Considering PSA Screening
Keywords: Prostate cancer; Decision support intervention (DESI); Shared medical appointments (SMA); Comparative effectiveness research (CER)
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Mail DVD (Experimental)
  Interventions: Behavioral: DESI for home viewing
- Invite to SMA to view and discuss DESI (Experimental)
  Interventions: Behavioral: DESI for viewing at Shared Medical Appointment
- SMA and DVD (Experimental)
  Interventions: Behavioral: Option of SMA and DESI or DESI only
- Encouraged to talk to physician (No Intervention)

INTERVENTIONS:
Behavioral: DESI for home viewing — Decision support intervention is a 31 minute DVD mailed to the patients in all of the experimental groups. The program explains the function and location of the prostate and the nature of prostate cancer, including its associated mortality. Next, the program describes the different tests that are used to detect prostate cancer including the digital rectal exam, prostate specific antigen (PSA) test and prostate biopsy.
  Arms: Mail DVD
Behavioral: DESI for viewing at Shared Medical Appointment — Shared medical appointment (SMA) sessions will be led by a mid-level provider. The sessions will begin with an introduction about the importance of making an informed decision about prostate cancer screening. The PSA decision support intervention will be shown and then, after the program, participants will be invited to ask questions or share their thoughts and feelings. At the end of the session, information on how to obtain a PSA screening test will be provided to participants. Men who decide in favor of a PSA test immediately following a SMA will be given a lab order which they can use to have the test performed.
  Arms: Invite to SMA to view and discuss DESI
Behavioral: Option of SMA and DESI or DESI only — Shared medical appointment (SMA) sessions will be led by a mid-level provider. The sessions will begin with an introduction about the importance of making an informed decision about prostate cancer screening. The PSA decision support intervention will be shown and then, after the program, participants will be invited to ask questions or share their thoughts and feelings. At the end of the session, information on how to obtain a PSA screening test will be provided to participants. Men who decide in favor of a PSA test immediately following a SMA will be given a lab order which they can use to have the test performed.
  Arms: SMA and DVD

SUMMARY:
In this study we will compare 3 strategies for systematic delivery of prostate cancer screening decision support interventions (DESI) to usual care and examine their impact on screening decisions and subsequent healthcare utilization using a randomized control design.

We hypothesize men who are given the opportunity to review a DESI by one of the 3 strategies will be less likely to opt for prostate cancer screening, and will have lower subsequent healthcare utilization than men in the control group.

DETAILED DESCRIPTION:
We will use a randomized experimental design to compare the effects of 3 different strategies to implement a prostate cancer screening decision support intervention (DESI) with a control condition in primary care in 2 clinical systems - PAMF (Palo Alto Medical Foundation) and UNC. The primary outcomes of interest are men's screening decisions and their subsequent healthcare utilization. Secondary outcomes include the likelihood that they review the DESI and their decision-specific knowledge. The 3 strategies selected by the PAMF and UNC health systems are: (1) mailing men a DESI in DVD; (2) inviting men to participate in a shared (group) medical appointment (SMA) to watch and discuss the DESI with a healthcare provider and other men; and (3) providing men options by inviting them to a SMA while also providing them a DESI in DVD which they can use individually if they are unable or choose not to attend a SMA. The 3 groups will be compared to a control condition that does not receive a DESI but will be encouraged to discuss prostate cancer screening with their physician. Because of its significantly larger patient population, the PAMF site will also evaluate these outcomes by targeting screening-naïve patients on their 50th birthday, when they first become guideline eligible to consider prostate cancer screening.

ELIGIBILITY:
Inclusion Criteria:

* age 50 or older
* do not have a prostate diagnosis
* have not had a PSA test in the past 10 months
* have not seen their primary care physicians in the last 3 months

Exclusion Criteria:

* Women

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2521 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
PSA test vs. No PSA test | 12 month follow-up
  We will determine whether a DESI viewing had an impact on testing.
Healthcare utilization and costs | 12 month follow-up
  All prostate specific health care utilization and cost will be estimate for each group.

SECONDARY OUTCOMES:
DESI viewing | 4 months after mailings
  Did the patient view the decision support intervention or not?
Decision specific knowledge | 4 months after mailings
  Patient's knowledge will be assessed with a validated 10-item measure.
Discussion with provider | 4 months after mailings
  Patients will be asked if they discussed prostate cancer screening with a healthcare provider.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen L Lewis, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill; Ming Tai-Seale, Ph.D, MPH, Principal Investigator — Palo Alto Medical Foundation
Locations (2):
- United States (2):
  - Palo Alto Medical Foundation Research Institute, Palo Alto, California
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina

REFERENCES:
- [Derived] Lewis CL, Adams J, Tai-Seale M, Huang Q, Knowles SB, Nielsen ME, Pignone MP, Walter LC, Frosch DL. A Randomized Controlled Effectiveness Trial for PSA Screening Decision Support Interventions in Two Primary Care Settings. J Gen Intern Med. 2015 Jun;30(6):810-6. doi: 10.1007/s11606-015-3214-9. Epub 2015 Feb 10. PMID 25666221